CLINICAL TRIAL: NCT01997970
Title: Non-exercise Activity Thermogenesis (NEAT) - Prevention and Treatment of Overweight and Obesity
Brief Title: NEAT - Prevention and Treatment of Overweight and Obesity.
Acronym: InphactUm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Tommy Olsson, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-338-31
Record Dates: First submitted 2013-11-02; First posted 2013-11-28 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Overweight; Obesity
Keywords: NEAT; Treadmill desk
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treadmill workstation (Experimental): Will receive a health talk with recommendations about diet and physical activity habits and will also receive a treadmill workstation at regular office site for 12 months.
  Interventions: Behavioral: Treadmill workstation; Behavioral: Health talk
- Control group (Experimental): Will receive a health talk with recommendations about diet and physical activity habits. Will continue to work with conventional office work at their regular desk.
  Interventions: Behavioral: Health talk

INTERVENTIONS:
Behavioral: Treadmill workstation — The intervention group will receive a treadmill workstation for 12 months. They will use this at self-selected speed and will be recommended to use this for at least 1 hour per day. Participants in the control group will continue with conventional office work at their regular desk. Participants in the intervention group will receive four boosting e-mails during the study period, in which they will be encouraged to use the treadmill.
  Arms: Treadmill workstation
Behavioral: Health talk — Participants in both groups will receive a health talk with recommendations about diet and physical activity habits.

SUMMARY:
This study will investigate the effect on Non-exercise Activity Thermogenesis (NEAT) when implementing active workstation at offices compared to conventional office work. The primary hypothesis is that this implementation will lead to a significant increase in time spent walking per day.

DETAILED DESCRIPTION:
NEAT consists of the energy expenditure of the physical activities that are non sporting-like and that we perform in our everyday life, such as walking, cleaning, shoveling snow etc. Which occupation we have play a big role in how much we are able to active our NEAT during our days and those who have more active jobs can expend up to 1500kcal more per day than those with sedentary jobs.

This study aims to try and increase NEAT at offices where sedentary time often is high. Participants will be randomized to either an intervention group or to a control group. Participants in the control group will continue to work at their regular desk, but will receive an individual health talk in the beginning of the study where diet and physical activity recommendations will be discussed.Participants in the intervention group will receive the same individual health talk and a treadmill desk, which they will use for 12 months at self-selected speed. They will be recommended to walk on the treadmill for at least 1 hour per day.

ELIGIBILITY:
Inclusion Criteria:

* Office workers with mainly sedentary tasks
* BMI 25-40

Exclusion Criteria:

* Severe depression and/or anxiety
* Exhaustion disorder
* Diabetes Mellitus
* Severe cardiovascular disease
* Severe kidney disease
* Musculoskeletal disorders that prohibit walking on a treadmill
* Contraindications for physical activity
* Thyroidea illness
* Pregnancy

For fMRI-study, additional exclusion criteria are:

* Implanted metal- or electrical devices
* Pregnancy
* Extraneous metal pieces in the body

Ages: 40 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity and sedentariness at 12 months | Baseline, 12 months
  Measured with an accelerometer (ActiGraph) and an inclinometer (ActivPAL).

SECONDARY OUTCOMES:
Change from baseline in metabolism at 12 months | Baseline, 12 months
  Metabolism: 2h glucose tolerance test. lipids, Hb1Ac
Change from baseline in anthropometrics at 12 months | Baseline, 12 months
  Length, height, weight, waist circumference, hip circumference, sagittal height, pulse, blood pressure.
Change from baseline in body composition at 12 months | Baseline, 12 months
  Measured with Dual X-Ray Absorptiometry (DXA)
Change from baseline in musculoskeletal pain at 12 months | Baseline, 12 months
  Measured with the Chronic Pain Grade Questionnaire
Change from baseline in stress at 12 months | Baseline, 12 months
  Measured by assessing cortisol levels in the saliva at 4 time points during one day. Also measured with the stress- and energy scale.
Change from baseline in depression/anxiety at 12 months | Baseline, 12 months
  Measured with the Hospital Anxiety and Depression Scale.
Change from baseline in Quality of Life at 12 months | Baseline, 12 months
  Measured with 2 questions from the SF-36.
Change from baseline in cognitive Function and functional brain response at 12 months | Baseline, 12 months
  Measured with a cognitive test battery and functional MRI (fMRI). Levels of Brain-Derived Neurotrophic Factor (BDNF) is measured in the plasma.
Qualitative interview study | 12 months
  Participants will be interviewed about experiences from being part of the study and about attitudes and factors that influences them to be physically active.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Olsson, Professor, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

REFERENCES:
- [Derived] Bergman F, Matsson-Frost T, Jonasson L, Chorell E, Sorlin A, Wennberg P, Ohberg F, Ryberg M, Levine JA, Olsson T, Boraxbekk CJ. Walking Time Is Associated With Hippocampal Volume in Overweight and Obese Office Workers. Front Hum Neurosci. 2020 Aug 20;14:307. doi: 10.3389/fnhum.2020.00307. eCollection 2020. PMID 32973475
- [Derived] Bergman F, Wahlstrom V, Stomby A, Otten J, Lanthen E, Renklint R, Waling M, Sorlin A, Boraxbekk CJ, Wennberg P, Ohberg F, Levine JA, Olsson T. Treadmill workstations in office workers who are overweight or obese: a randomised controlled trial. Lancet Public Health. 2018 Nov;3(11):e523-e535. doi: 10.1016/S2468-2667(18)30163-4. Epub 2018 Oct 12. PMID 30322782
- [Derived] Bergman F, Boraxbekk CJ, Wennberg P, Sorlin A, Olsson T. Increasing physical activity in office workers--the Inphact Treadmill study; a study protocol for a 13-month randomized controlled trial of treadmill workstations. BMC Public Health. 2015 Jul 10;15:632. doi: 10.1186/s12889-015-2017-6. PMID 26160221